CLINICAL TRIAL: NCT04782206
Title: the Added Analgesic Effect of S3 Root Pulsed Radiofrequency to Superior Hypogastric Plexus Block in Pelvic Cancer Pain. a Controlled, Randomized Study
Brief Title: S3 Root Pulsed Radiofrequency Added to Superior Hypogstric Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Assisstant Professor of Anesthesia, ICU, and Pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 366
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Pain Cancer; Pain, Chronic
Keywords: pelvic cancer pain; superior hypogastric plexus block; pulsed radiofrequency
MeSH Terms: conditions — Cancer Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): superior hypogastric plexus block
  Interventions: Procedure: superior hypogastric plexus block
- group 2 (Active Comparator): pulsed radiofrequency at S3 nerve root + superior hypogastric plexus block
  Interventions: Procedure: pulsed radiofrequency at S3 root plus superior hypogastric plexus block

INTERVENTIONS:
Procedure: superior hypogastric plexus block — superior hypogastric plexus chemical neurolysis
  Arms: group 1
Procedure: pulsed radiofrequency at S3 root plus superior hypogastric plexus block — pulsed radiofrequency neuromodulation at S3 root plus superior hypogastric plexus chemical neurolysis
  Arms: group 2

SUMMARY:
The investigators hypothesis that adding pulsed radiofrequency neuromodulation at S3 nerve root to superior hypogastric plexus chemical neurolysis improves analgesia in patients with chronic pelvic cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* pelvic cancer patients
* with pelvic pain not responding to oral analgesic medications
* side effects of oral analgesic medications

Exclusion Criteria:

* patients with metastatic cancer disease
* patients with significantly impaired organ functions
* patients with bleeding diathesis
* patients with mental disabilities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | from 30 min. after procedure to 2 months after it
  Visual Analogue Scale post-procedure

SECONDARY OUTCOMES:
complications | during the block procedure and within the first 24 hours after the block
  including transient paresthesia, rectal puncture, vascular penetration of one of the pelvic vessels, hematoma, infection, dural puncture, bowel/bladder dysfunction, pain on injection, hypotension from the sympathetic block or any other complication
procedure time | during the block procedure
  The time required to perform the block
Total oral analgesic consumption | in the first 24 hours after procedures and at 1,2,4 weeks and 2 months visits after it
  total MST consumption